CLINICAL TRIAL: NCT05060211
Title: Correlation Between Brain Lesion and Continence in Children with Cerebral Palsy: an Anatomical MRI Study
Brief Title: Incontinence and MRI Results in Children with Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702021000735
Record Dates: First submitted 2021-08-16; First posted 2021-09-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy; Lower Urinary Tract Symptoms
Keywords: cerebral palsy; lower urinary tract symptoms; Magnetic resonance imaging; brain lesion; incontinence
MeSH Terms: conditions — Cerebral Palsy; Lower Urinary Tract Symptoms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Vancouver symptom score for dysfunctional elimination syndroms — Validated questionnaire concerning bladder and bowel symptoms
  Other Names: VSSDES
Other: Magnetic resonance imaging — Known MRI results of the patient file
  Other Names: MRI

SUMMARY:
More than 50 % of children and adults with cerebral palsy experience lower urinary tract symptoms (LUTS). This can negatively influence quality of life of the child and the total social environment.

Previous research demonstrated that the brain lesion, characteristic for cerebral palsy (CP), is a prognostic factor for the functional abilities of a child with CP. Previous research within our department demonstrated functional impairment as a risk factor for incontinence. This demonstrates an indirect connection between the brain lesion and incontinence of a child with CP. However, this connection isn't alway correct as some children with high functionality also demonstrate incontinence.

As bladder control is also regulated by higher brain centers, the present study wants to investigate a direct connection between the brain lesion of the child, visible by means of MRI, and the incontinence status of the child. .

DETAILED DESCRIPTION:
The current study is a cross-sectional observational study in which a correlation is investigated between known anatomical MRI results and the continence status of a child with CP.

Although neuroimaging isn't seen as a requirement for the definition and diagnosis of CP2, MRI imaging is often part of diagnostic evaluation. The Surveillance of Cerebral Palsy in Europe (SCPE) working group composed the MRI classification system or MRICS classifying neuroimaging results in maldevelopments, predominant white matter injury, predominant grey matter injury, miscellaneous and normal. These results will be correlated with results of the validated Vancouver symptoms score for dysfunctional elimination syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* MRI investigation in history
* Dutch or French speaking child and parent

Exclusion Criteria:

* No MRI investigation in history
* Child or parent not speaking Dutch or French

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy attending yearly or half yearly follow-up consultation
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incontinence ratio | During cross-sectional testing
  Amount of patients with incontinence in the different MRICS-groups (MRI classification system for children with CP).

SECONDARY OUTCOMES:
Amount of Lower urinary tract symptoms in different MRICS-groups | During cross-sectional testing
  Score of 'Vancouver symptom score for dysfunctional elimination syndrome'-questionnaire and individual questions in the different MRICS- groups (MRI classification system for children with CP).
Amount of bladder symptoms in different MRICS-groups | During cross-sectional testing
  Score of individual questions from the 'Vancouver symptom score for dysfunctional elimination syndrome' questionnaire in the different MRICS- groups (MRI classification system for children with CP).

CONTACTS AND LOCATIONS:
Overall Officials: Bieke Samijn, dr., Principal Investigator — Ghent University Hospital/Ghent University
Locations (1):
- Ghent University Hospital, Ghent, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No